CLINICAL TRIAL: NCT03850366
Title: HLA-Haploidentical Peripheral Blood Stem Cell Transplantation With Post-transplant Cyclophosphamide and Bortezomib Following Fludarbine/Melphalan/Total Body Irradiation Conditioning Regimen
Brief Title: HLA-Haploidentical Peripheral Blood Stem Cell Transplantation With Post-transplant Cyclophosphamide and Bortezomib
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Henry Ford Health System (Other)
Responsible Party: Principal Investigator, Shatha Farhan, Principal Investigator, Henry Ford Health System
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 10313
Record Dates: First submitted 2019-02-20; First posted 2019-02-21 (Actual); Last update posted 2025-02-11 (Actual); Status verified 2025-02

CONDITIONS: Hematological Malignancy
MeSH Terms: conditions — Hematologic Neoplasms | interventions — Bortezomib; Cyclophosphamide

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Bortezomib (Experimental)
  Interventions: Drug: Bortezomib

INTERVENTIONS:
Drug: Bortezomib — GVHD prophylaxis
  Other Names: cyclophosphamide

SUMMARY:
Now haplo stem cell transplant using bone marrow or peripheral blood is becoming more feasible with better regimens to prevent graft versus host disease (GVHD) like post transplant cyclophosphamide , tacrolimus, mycophenolate . Recently Bortezomib has also been shown to inhibit dendritic cells maturation and function and possesses a number of other favorable immunomodulatory effect that can prevent GVHD and help enhance immune reconstitution. this study is to assess the engraftment rate in patients with hematologic malignancies who need allogeneic stem cell transplant but do not have a suitable matched related or unrelated stem cell donor and will get T-cell replete HLA-Haploidentical allogeneic peripheral stem cell transplantation using post transplant Cyclophosphamide and bortezomib

ELIGIBILITY:
Inclusion Criteria:

* 18-65 years old patient lacking a matched related donor or unrelated donor but have a related haploidentical donor (</= 7/8 allele match at the A, B, C, DR loci with a minimum match of 5/10 is required) is identified
* Candidate for stem cell transplant in a malignant hematological condition
* Karnofsky Performance Scale 0-1
* Available donor able to undergo a Peripheral blood stem cells collection
* Bilirubin </= 1.5 mg/dl , aspartate aminotransferase (AST) or alanine aminotransferase (ALT) </= 200 IU/ml for adults.
* Serum creatinine clearance >/=60 ml/min (calculated with Cockroft-Gault formula)
* Diffusing capacity for carbon monoxide (DLCO) >/= 45% predicted corrected for hemoglobin.
* Left ventricle ejection fraction > 40%.
* Patient or patient's legal representative, parent(s) or guardian should provide written informed consent.

Exclusion Criteria:

* Adult who has a suitable related or unrelated donor or cord units available for transplant. Suitable donors include 8/8 (HLA-A,B,C and DR, with all loci high-resolution typing) or 7/8 related or unrelated donor available within 42 days of search initiation
* HIV positive; active hepatitis B or C
* Patients with active uncontrolled infections.
* Liver cirrhosis
* Uncontrolled central nervous system involvement by tumor cells
* Positive Beta Human chorionic gonadotropin (HCG) test in a woman with child bearing potential defined as not post-menopausal for 12 months or no previous surgical sterilization.
* Inability to comply with medical therapy or follow-up

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2016-03-08 (Actual); Primary Completion 2027-01-01 (Estimated); Study Completion 2027-01-01 (Estimated)

PRIMARY OUTCOMES:
engraftment rate | within 30 days post transplant
  rate of neutrophil and platelet engraftment post stem cell transplant

CONTACTS AND LOCATIONS:
Locations (1):
- Henry Ford hospital, Detroit, Michigan, United States